CLINICAL TRIAL: NCT00477061
Title: Double Blind Randomized Study of Morphine Analgesia in Patients With Acute Appendicitis
Brief Title: Morphine Analgesia in Patients With Acute Appendicitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AG11
Record Dates: First submitted 2007-05-20; First posted 2007-05-22 (Estimated); Last update posted 2007-05-22 (Estimated); Status verified 2007-05

CONDITIONS: Appendicitis
Keywords: MORPHINE; ANALGESIA; ACUTE APPENDICITS
MeSH Terms: conditions — Appendicitis; Agnosia | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Morphine

SUMMARY:
The purpose of the study is to evaluate morphine effect on pain reduction and diagnostic accuracy in patients admitted to emergency ward with the diagnosis of acute appendicitis.

DETAILED DESCRIPTION:
Analgesic administration for pain control in patients with acute abdominal pain, regarding acute appendicitis, is controversial. Despite the results previous studies indicating the safeness of analgesic use in ED for acute abdominal pain, physicians still prefer to postpone their use after performing surgical evaluations. Since many patients admitted to ED are unlikely to receive prompt surgical consultation, many of them need pain relief to prevent unnecessary suffering. On the other hand such pain relief must not interfere with the diagnosis and treatment of patients and do not cause any complications. Morphine is a common and effective analgesic which, if shown to have no effect on correct diagnosis of acute abdomen, can be used for this purpose.

Thus we evaluated morphine effect on pain reduction and diagnostic accuracy in patients admitted to ED with the diagnosis of acute appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* clinical signs of acute appendicitis
* planned for appendectomy
* supposed to wait for at least 1 hour in the ED before operation

Exclusion Criteria:

* suspicion to perforated appendicitis
* being under the age of 13
* pregnancy (according to history and ß-HCG result)
* opium addiction
* systolic blood pressure of less than 90 mmHG
* known cases of chronic obstructive pulmonary disease (COPD)
* known sensitivity to morphine
* history of sickle cell disease
* self administration of analgesics before enrollment
* refusal to participate

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2004-01; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Pain Intensity

SECONDARY OUTCOMES:
Diagnostic Accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Asieh Golozar, MD, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Sina General Hospital, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Amoli HA, Golozar A, Keshavarzi S, Tavakoli H, Yaghoobi A. Morphine analgesia in patients with acute appendicitis: a randomised double-blind clinical trial. Emerg Med J. 2008 Sep;25(9):586-9. doi: 10.1136/emj.2007.050914. PMID 18723709